CLINICAL TRIAL: NCT03099915
Title: Asthma Attack in the Emergency Department : Reasons Of This Attendance
Acronym: AERO
Status: Completed | Type: Observational
Sponsor: Olivier CHASSANY (Other)
Collaborators: EA 7334, Patient-Centered Outcomes Research (Unknown); Bichat Hospital (Other); Beaujon Hospital (Other)
Responsible Party: Sponsor-Investigator, Olivier CHASSANY, Director, University Paris 7 - Denis Diderot
Organization: University Paris 7 - Denis Diderot (Other)
Other Study IDs: AERO
Record Dates: First submitted 2017-03-17; First posted 2017-04-04 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Asthma Attack; Emergency Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: completion of self-reported questionnaires — Single completion: Participants will have to complete self-reported questionnaires based on gina criteria and 12-item general health questionnaire

SUMMARY:
Objective: Identify modifiable factors that may affect asthma control and the use of emergency room to define customized interventions for the management of asthma prior to emergency room.

Emergency department attendance is always a sign of poor balance or control of asthma. In spite of a decrease in the number of deaths that has been halved in 20 years and hospitalization due to asthmatic disease, the use of emergency center for this disease has not decreased. We now know that the passage through emergencies and hospitalization for aggravation of asthma is in itself a factor of mortality. Acting on the determinants of poor balance or control of asthma is essential to further reduce the mortality and morbidity of asthma.

DETAILED DESCRIPTION:
There is two parts in this study:

Part 1 - Qualitative study by individual interviews until data saturation (although about ten patients should be enough to capture the concepts of interest) on the factors that induce an imbalance of asthma (based on the GINA (Global Initiative for Asthma) report whose criteria are validated).

An interview guide will be written to systematically address all aspects related to asthma control.

In agreement with the patient the interview will be recorded, and the verbatim will be transcribed and coded using a software (Nvivo version 10).

Preparation of a questionnaire

A questionnaire will be developed from:

* analysis of patient verbatim
* other data: GINA criteria, psychological criteria (psychological distress is assessed by the 12-item general health questionnaire (GHQ-12) which is valid psychometric tools in French) and social criteria.

Part 2-Observational cohort qualitative study. The questionnaire thus prepared will be placed in the patient file upon admission. As soon as possible it will be filled by the patient after improvement of his condition and collected by the doctor or nurse who took care of the patient.

To obtain sufficient power to demonstrate significant associations, and assuming that 15 variables are taken into account in a multivariate model and based on the recommendations of 10 subjects per variable, 150 patients are required.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Ambulatory patient, visiting one of these centers
* Diagnosis of asthma already evolving for more than 6 months
* Prescription of treatment for more than 3 months
* Patient who can read and write French
* Agreement for an individual interview (Part 1) or fill up a self-questionnaire (Part 2)
* Health insurance coverage

Exclusion Criteria:

* Patients with other etiology that may explain their dyspnea: heart failure, chronic obstructive pulmonary disease , pneumopathy
* Patients with a social background that is not compatible with the study: a patient who does not speak French, is homeless or does not have a telephone number
* Inpatients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults visiting emergency department for asthma attack
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Poor observance of GINA criteria | Less than 24 hours: the outcome measure will be assessed the visiting day at emergency room, when the asthma attack will be solved, before discharge from hospital
  Explanation of Asthma imbalance by poor observance and knowledge of GINA global strategy for asthma management and prevention criteria.

SECONDARY OUTCOMES:
GHQ-12 Psychometric tool | Less than 24 hours: the outcome measure will be assessed the visiting day at emergency room, when the asthma attack will be solved, before discharge from hospital
  Psychological distress caused by asthma will be measured by general health questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CHASSANY, MD, PhD, Study Director — EA 7334, University Paris-Diderot, Paris; Prabakar VAITTINADA AYAR, MD, Principal Investigator — Hôpital Bichat-Claude Bernard; Enrique CASALINO, MD, Study Chair — Hôpital Bichat-Claude Bernard
Locations (2):
- France (2):
  - Service d'accueil des urgences Hôpital Beaujon, Clichy
  - Service d'acceuil des urgences hôpital Bichat- Claude Bernard, Paris

IPD SHARING:
Plan to Share IPD: No